CLINICAL TRIAL: NCT00564954
Title: A Randomized, Multi-center, Double-blind, Cross-over Study Comparing the Efficacy and Safety of Focalin® XR 20 mg Versus Placebo at the 0.5 Hour Timepoint (Post-dose) in Children (6-12 Years) With Attention-Deficit/Hyperactivity Disorder (ADHD) in a Laboratory Classroom Setting
Brief Title: A Study of Dex-methylphenidate Extended Release in Children (6-12 Years) With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRIT124EUS19
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Results first posted 2009-03-30 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; children; laboratory classroom; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dexmethylphenidate Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Dex-methylphenidate hydrochloride (Focalin XR) (Experimental): 20 mg capsule orally once a day for 7 days
  Interventions: Drug: Dex-methylphenidate hydrochloride extended-release (Focalin XR)
- Placebo (Placebo Comparator): orally once a day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dex-methylphenidate hydrochloride extended-release (Focalin XR) — 20 mg capsule orally once a day for 7 days
  Other Names: Focalin XR
  Arms: Dex-methylphenidate hydrochloride (Focalin XR)
Drug: Placebo — orally once a day for 7 days
  Arms: Placebo

SUMMARY:
This study compared the efficacy of dex-methylphenidate extended release 20 mg versus placebo during an 8-hour laboratory classroom day.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 6-12 years, inclusive.
* Subjects meeting the DSM-IV criteria for ADHD of any type, as established by the K-SADS-PL (Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime Version). If a DSM-IV-defined ADHD diagnosis is difficult to establish due to possible co-morbidity, the subject will not be enrolled into the study.
* Subjects should be on a stabilized total daily dose or nearest equivalent of 40-60 mg methylphenidate or 20-30 mg of d-methylphenidate for at least two weeks prior to screening visit (Concerta® 36 mg and 54 mg is allowable)

Exclusion Criteria:

* Parent or guardian unable or unwilling to complete the Conner's ADHD/DSM-IV Scale for Parents (CADS-P) and the Daily Diary Card
* Diagnosed with a tic disorder or Tourette's syndrome
* History of seizure disorder
* The presence of a known medical condition that would preclude the use of methylphenidate. A history (within the past year) or presence of clinically significant cardiovascular, cerebrovascular, renal, hepatic, gastrointestinal, pulmonary, immunological, hematological, endocrine, or neurological disease
* ALT, AST, GGPT or serum creatinine greater then 2X the ULN at Screening
* A history of psychiatric illness or substance use disorder (e.g., schizophrenia, bipolar disorder, autism, abuse or dependence, depression, severe Conduct Disorder or severe Oppositional defiant disorder)
* Subjects who have participated in an investigational trial within the past 4 weeks (28 days) are excluded
* Subjects who are currently taking antidepressants or other psychotropic medication
* Subjects who have initiated psychotherapy during the three months prior to randomization
* Subjects with a positive urine drug screen
* Subjects who have a history of poor response or intolerance to methylphenidate or d-methylphenidate

Other protocol defined inclusion/exclusion criteria may apply

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lubbock, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Dex-methylphenidate Hydrochloride (Focalin XR) Then Placebo: Period 1: One 20 mg capsule of Focalin XR taken once daily in the morning for one week followed by Period 2: one week of placebo taken once daily in the morning.
- Placebo Then Dex-methylphenidate Hydrochloride (Focalin XR): Period 1: One week of placebo taken once daily in the morning followed by Period 2: one week of one 20 mg capsule of Focalin XR taken once daily in the morning.
Period: Period 1- 1 Week
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) Then Placebo | Placebo Then Dex-methylphenidate Hydrochloride (Focalin XR)
Started | 44 | 42
Completed | 44 | 42
Not Completed | 0 | 0
Period: Period 2- 1 Week
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) Then Placebo | Placebo Then Dex-methylphenidate Hydrochloride (Focalin XR)
Started | 44 | 42
Completed | 44 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) Then Placebo | Placebo Then Dex-methylphenidate Hydrochloride (Focalin XR) | Total
Number analyzed (Participants) | 44 | 42 | 86
Age Continuous [Mean (Standard Deviation); unit: years] | 9.5 (2.0) | 9.4 (1.4) | 9.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 28 | 25 | 53

OUTCOME MEASURES:

1. Secondary Outcome: Change From Pre-dose (0 hr) in SKAMP Combined Score at All Times Excluding the 0.5 Hour Timepoint (Hours 1, 2, 4, 6, 8)
Description: SKAMP rating scale is comprised of 13 questions (7 questions on attention and 6 questions on deportment) evaluating classroom behavior; answers to each question range from 0 (normal, no impairment) to 6 (maximum impairment) for a total possible combined score of 0 to 78.
Time Frame: 0, 1, 2, 4, 6, and 8 hr
Population: Intent to Treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Dex-methylphenidate Hydrochloride (Focalin XR): Summary of the one week treatment on dex-methylphenidate hydrochloride (Focalin XR), 20 mg capsule orally once a day, for all 86 patients regardless of sequence.
- Placebo: Summary of the one week treatment on placebo once a day orally for 7 days for all 86 patients regardless of sequence.
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) | Placebo
Number analyzed (Participants) | 86 | 86
score on a scale
  1 hour | -6.358 (0.993) | 5.670 (0.991)
  2 hours | -11.573 (0.856) | 5.467 (0.854)
  4 hours | -11.395 (0.847) | 3.925 (0.844)
  6 hours | -10.622 (0.950) | 5.346 (0.952)
  8 hours | -10.260 (0.988) | 3.621 (0.986)

2. Secondary Outcome: Change From Pre-dose in SKAMP Attention Score at All Timepoints (0.5, 1, 2, 4, 6, 8)
Description: SKAMP attention sub-scale is comprised of 7 questions evaluating concentration in the classroom; answers to each question range from 0 (normal, no impairment) to 6 (maximum impairment) for a total possible combined score of 0 to 42.
Time Frame: 0, 0.5, 1, 2, 4, 6, and 8 hours
Population: Intent to Treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) | Placebo
Number analyzed (Participants) | 86 | 86
score on a scale
  0.5 hour | -0.825 (0.524) | 0.862 (0.520)
  1 hour | -4.208 (0.589) | 2.304 (0.584)
  2 hours | -6.591 (0.507) | 2.465 (0.504)
  4 hours | -6.722 (0.506) | 1.183 (0.503)
  6 hours | -5.819 (0.582) | 2.715 (0.580)
  8 hours | -6.061 (0.584) | 1.415 (0.580)

3. Secondary Outcome: Change From Pre-dose in SKAMP Deportment Score
Description: SKAMP deportment sub-scale is comprised of 6 questions on behavior in the classroom; answers to each question range from 0 (normal, no impairment) to 6 (maximum impairment) for a total possible combined score of 0 to 36.
Time Frame: 0, 0.5, 1, 2, 4, 6 and 8 hours
Population: Intent to Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) | Placebo
Number analyzed (Participants) | 86 | 86
score on a scale
  0.5 hour | 0.127 (0.550) | 2.226 (0.550)
  1 hour | -1.863 (0.564) | 3.103 (0.564)
  2 hours | -4.850 (0.499) | 2.881 (0.499)
  4 hours | -4.420 (0.526) | 2.511 (0.526)
  6 hours | -4.614 (0.541) | 2.393 (0.541)
  8 hours | -3.939 (0.560) | 1.969 (0.560)

4. Secondary Outcome: Change From Pre-dose (0 hr.) in Permanent Product Measure of Performance (PERMP) Math Test-Attempted Scores at All Timepoints (0.5, 1, 2, 4, 6, 8)
Description: Number of math questions attempted within a 10 minute period.
Time Frame: 0, 0.5, 1, 2, 4, 6 and 8 hours
Population: Intent to Treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: questions attempted
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) | Placebo
Number analyzed (Participants) | 86 | 86
questions attempted
  0.5 hour | 6.93 (2.96) | -4.74 (2.96)
  1 hour | 33.26 (3.66) | -12.18 (3.66)
  2 hours | 45.52 (3.61) | -10.19 (3.61)
  4 hours | 45.01 (3.60) | -7.42 (3.60)
  6 hours | 37.33 (3.82) | -16.70 (3.84)
  8 hours | 44.04 (3.50) | -10.08 (3.50)

5. Secondary Outcome: Change From Pre-dose in Number of Math Questions Answered Correctly on the Permanent Product Measure of Performance (PERMP) Math Test
Description: Number of math questions answered correctly within a 10 minute period.
Time Frame: 0, 0.5, 1, 2, 4, 6 and 8 hours
Population: Intent to Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: questions correct
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) | Placebo
Number analyzed (Participants) | 86 | 86
questions correct
  0.5 hour | 7.10 (2.72) | -5.96 (2.72)
  1 hour | 31.10 (3.34) | -13.21 (3.34)
  2 hours | 44.92 (3.44) | -11.09 (3.44)
  4 hours | 43.64 (3.37) | -7.52 (3.37)
  6 hours | 37.78 (3.55) | -16.90 (3.57)
  8 hours | 43.37 (3.40) | -11.44 (3.40)

6. Primary Outcome: Change From Pre-dose (0 hr [Hour]) on the Swanson, Kotkin, Agler, M-Flynn & Pelham (SKAMP) Rating Scale Combined Score at 0.5 Hour During the 8- Hour Laboratory Classroom Day
Description: as for outcome 1
Time Frame: 0 hr and 0.5 hr post-dose
Population: Intent to Treat (ITT) population: All randomized patients who had at least one dose of study medication and who had at least one post-dose efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) | Placebo
Number analyzed (Participants) | 86 | 86
score on a scale | -0.969 (0.909) | 3.336 (0.907)

ADVERSE EVENTS:
Arm/Group | Dex-methylphenidate Hydrochloride (Focalin XR) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary; however, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.